CLINICAL TRIAL: NCT03130088
Title: European Registry of Cardiac Arrest - Study Two (EuReCa TWO) An International, Prospective, Multi-centre, Three-month Survey of Epidemiology, Treatment and Outcome of Patients Suffering an Out-of-hospital Cardiac Arrest in Europe
Brief Title: European Registry of Cardiac Arrest Study Two
Acronym: EuReCa TWO
Status: Completed | Type: Observational
Sponsor: German Resuscitation Registry (Other)
Responsible Party: Sponsor
Other Study IDs: EuReCa TWO
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Resuscitation Registry
Keywords: Out-Of-Hospital Cardiac Arrest; Resuscitation Registry; EuReCa TWO
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention planed — no intervention planed

SUMMARY:
This study will evaluated the epidemiology and the outcome of patients suffering out-of-hospital cardiac arrest in 27 european nations. The special focus in the EuReCa TWO study is on bystander CPR.

DETAILED DESCRIPTION:
The importance of the establishment of out-of-hospital cardiac arrest (OHCA) registries as a critical step in improving OHCA outcomes is recognised from clinical, academic and political perspectives 1-4. The aim of the EuReCa project is to establish a European Registry of Cardiac Arrest to provide quality benchmarking for OHCA measurement in Europe based on Utstein style data collection, so that variations in OHCA incidence, management and outcomes can be identified 5,6.

The EuReCa ONE project secured the collaboration of 27 European countries. During October 2014, data was collected from each of these countries, resulting in the most comprehensive estimate of OHCA incidence and outcomes to date 7. As expected, the proportion of variation between data collection from individual countries was considerable. While much of this variation is likely to be attributable to patient and system level differences, some variation was a consequence of the difference in proportions of countries covered by data collection, and may also have been caused by differences in how key variables were interpreted.

Improving data quality is an incremental process therefore in EuReCa TWO, we aim to build on the work of EuReCa ONE and further improve understanding of OHCA incidence, management and outcome across the continent. Key to the overall aim of achieving quality benchmarking is to ensure that EuReCa data collection is comprehensive and reliable.

Essential to the aims of the EuReCa project is that the data collected on each link of the Chain of Survival is comparable across participating countries. During EuReCa ONE, it was noted that the term 'bystander CPR' was interpreted differently across countries. A subsequent European survey of interpretation of the term 'bystander' and 'bystander CPR' confirmed this observation.

In order to enhance the key quality requirements of comprehensiveness and reliability, the aims of the EuReCa TWO project will be as follows:

* Expand the EuReCa network
* Improve the understanding of the role of bystanders in OHCA in Europe

In order to achieve these aims, the following objectives will be fulfilled:

* Encourage participating countries to aim for national data collection and encourage additional countries to participate
* In order to provide more robust estimates of incidence, management and outcome, increase the data collection period, increase the period of data collection to three months (1st October to 31st December 2017)
* Identify consistency and variation in the use of the term 'bystander CPR'
* Describe the incidence of 'bystander CPR' and its influence on OHCA outcome

EuReCa TWO is expected to result in the creation of the largest ever database of OHCA European data, which has been collected over a single time period, using consistent data definitions. This will provide the opportunity to generate more robust estimates of OHCA incidence and outcome for particular subgroups.

2. Research Questions

In order to build on previous work and improve the robustness of estimates, the Research Questions in EuReCa TWO will closely mirror those of EuReCa ONE:

* What proportion of each country's national population is covered by data collection?
* What is the incidence of confirmed OHCA attended by the EMS in different European regions?
* What is the incidence of any CPR (cardiopulmonary resuscitation) attempted in OHCA throughout Europe?
* What proportion of CPR is started by:

  * Bystander - on scene by chance
  * Person alerted to scene by ambulance dispatch
  * EMS?
* What is the age and gender profile of those who provide CPR before EMS arrival?
* In OHCA, what is the initial cardiac arrest rhythm of the patients where bystanders or EMS starts CPR or any other resuscitation intervention - shockable or non-shockable?
* In patients where CPR was started by bystanders or EMS, what is the incidence and rate of any return of spontaneous circulation (ROSC) after out-of-hospital cardiac arrest?
* What is the incidence of patients never transported due to being declared dead on scene?
* What is the patient status at handover from EMS to emergency department or hospital system with ongoing additional treatment in the next step of care (ROSC, ongoing CPR, dead)?
* What is the incidence of patients who are still alive 30 days (whether in-hospital or discharged) after their cardiac arrest event and/or what is the incidence of patients who are discharged alive from hospital?
* In patients with a witnessed collapse (witnessed by bystanders and/or EMS), found in a shockable rhythm and with an event of medical aetiology (i.e. Utstein comparator group):

  * What is the incidence of ROSC at hospital admission (at time of being handed over from EMS to emergency department or hospital system with ongoing additional treatment e.g. PCI) for the Utstein group
  * What is the incidence of patients who are still alive at 30 days (whether in-hospital or discharged) after their cardiac arrest event and/or what is the incidence of patients who are discharged alive from hospital in the Utstein group?
* What factors determine ROSC, admission and survival (as defined in questions above)?

Secondary Research Questions

* What is the European incidence of and percentage survival from OHCA with a traumatic aetiology?
* What is the European incidence of and percentage survival from OHCA in cases brought to hospital with unsustained ROSC and/or ongoing CPR?

ELIGIBILITY:
Inclusion Criteria:

* All patients who suffer an out of hospital cardiac arrest * and are attended by the EMS at any stage during the event. This study will include all events that occur between 00:00 on 1st October 2017 and 23:59 on 31st December 2017. Patients will be included irrespective of their age, gender or personal factors.

These inclusion criteria include all patients who receive resuscitation (chest compression and/or defibrillation of any type)

* By the EMS
* Before the arrival of the EMS with continued resuscitation by the EMS
* Before the arrival of the EMS, that is immediately stopped (for any reason) when the EMS arrives
* Patients who achieve ROSC before the arrival of the EMS It also includes patients found or declared dead (for any reason). Some countries or registries may not be able to provide all necessary data to answer every research question. These registries will not be included in the analysis of the related research questions.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population in the 27 participatiing nations, suffering out-of-hospital cardiac arrest and are treated/attended by the EMS
Sampling Method: Probability Sample
Enrollment: 35000 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
ROSC | latest inclusion December, 31st 2017
  return of any circulation after out-of-hopsital cardiac arrest

SECONDARY OUTCOMES:
30 day survival | 30 days, latest inclusion January, 31st 2018
  status of survival after 30 days after out-of-hospital cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Thorsten Graesner, MD, Principal Investigator — University Hospital Schleswig-Holstein, Department of Anaesthesiology and Intensive Care Medicine, Kiel, Germany
Locations (1):
- Germany ans 26 other european registries, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zadlo A, Bednarek-Chaluda M, Karpinska IA, Cebula G, Tokarek T; www.linkedin.com/in/anna-zadlo230789. Association between time of day and outcomes after out-of-hospital cardiac arrest in Poland: an analysis of the EuReCa registry. BMJ Open. 2025 Oct 20;15(10):e105187. doi: 10.1136/bmjopen-2025-105187. PMID 41120136
- See also: Related Info — http://www.eureca-two.eu